CLINICAL TRIAL: NCT04080921
Title: The Outcomes of Autologous Bone Marrow-derived Mononuclear Cell Transplantation In-patient With Neurological Sequelae Due to Encephalitis or Meningitis at Vinmec International Hospital
Brief Title: Stem Cell Transplantation In-patient With Neurological Sequelae Due to Encephalitis or Meningitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS. ĐT.19H2
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Encephalitis; Meningitis
Keywords: encephalitis; meningitis; neurological sequelae due
MeSH Terms: conditions — Encephalitis; Meningitis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cell transplantation (Experimental): Stem cell transplantation 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 6 months afterward
  Interventions: Combination Product: Stem cell transplantation

INTERVENTIONS:
Combination Product: Stem cell transplantation — Transplantation of Autologous Bone Marrow Mononuclear Cells

SUMMARY:
To evaluate the safety and efficacy of autologous bone marrow-derived mononuclear cell transplantation in-patient with neurological sequelae due to encephalitis or meningitis

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of autologous bone marrow-derived mononuclear cell in 22 patients with neurological sequelae due to encephalitis or meningitis at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

* Neurological sequelae due to encephalitis or meningitis

Exclusion Criteria:

* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Total Score of Gross Motor Function Measure (GMFM-88) | Baseline, 6 months, and 12 months after transplantation
  The Gross Motor Function Measure - 88 items (GMFM-88) is a standardized observational tool used to evaluate changes in gross motor function in children with cerebral palsy and other disabilities. The total score ranges from 0 to 264, with higher scores representing better gross motor function
Change in Muscle Tone Assessed by Modified Ashworth Scale (MAS) | Baseline, 6 months, and 12 months after transplantation
  The Modified Ashworth Scale (MAS) is a clinical tool used to measure muscle tone and the degree of spasticity in patients with neurological conditions. The scale ranges from 0 to 4, with an additional 1+ category. Scores are interpreted as follows: 0 indicates no increase in muscle tone, 1 indicates a slight increase in muscle tone with a catch and release, 1+ indicates a slight increase with minimal resistance throughout the remainder of the range of motion, 2 indicates a more marked increase in muscle tone through most of the range of motion, 3 indicates considerable increase in muscle tone making passive movement difficult, and 4 indicates that the affected part(s) are rigid in flexion or extension. Lower scores represent better outcomes (normal muscle tone), while higher scores represent worse outcomes

SECONDARY OUTCOMES:
Number of adverse events | Through study completion, an average of 12 months
  Examples of adverse events to look for: fever, infections, vomit, epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bansal H, Singh L, Verma P, Agrawal A, Leon J, Sundell IB, Koka PS. Administration of Autologous Bone Marrow-Derived Stem Cells for Treatment of Cerebral Palsy Patients: A Proof of Concept. J Stem Cells. 2016;11(1):37-49. PMID 28296863
- [Result] Nguyen LT, Nguyen AT, Vu CD, Ngo DV, Bui AV. Outcomes of autologous bone marrow mononuclear cells for cerebral palsy: an open label uncontrolled clinical trial. BMC Pediatr. 2017 Apr 12;17(1):104. doi: 10.1186/s12887-017-0859-z. PMID 28403842